CLINICAL TRIAL: NCT00365690
Title: Telephone-Delivered Coping Improvement Intervention for HIV Infected Older Adults
Brief Title: Effectiveness of a Telephone-Delivered Behavioral Treatment to Improve the Quality of Life of Older Adults With HIV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH078749 (NIH); R01MH078749 (NIH); DAHBR ASNM
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2013-05

CONDITIONS: HIV Infections; Depression
Keywords: AIDS; Older Adults; Telephone; Telemedicine
MeSH Terms: conditions — HIV Infections; Depression; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Participants will receive individual therapy upon request
  Interventions: Behavioral: Individual therapy
- 2 (Active Comparator): Participants will receive telephone-administered supportive-expressive group therapy
  Interventions: Behavioral: Telephone-administered supportive-expressive therapy
- 3 (Experimental): Participants will receive telephone-administered coping improvement group therapy
  Interventions: Behavioral: Telephone-administered coping improvement therapy

INTERVENTIONS:
Behavioral: Telephone-administered coping improvement therapy — Telephone-administered coping improvement therapy is aimed to improve coping in older adults living with HIV/AIDS. Participants will partake in 12 weekly conference calls lasting approximately 90 minutes each. Six to eight participants and two group facilitators will be connected via telephone each week. Separate conference call groups will be conducted for men who have sex with men, heterosexual men, and women. Cognitive behavioral principles will be used to evaluate stressor severity, develop problem- and emotion-focused coping skills, determine the relationship between coping strategies and stressor controllability, and optimize coping through use of social support resources. Between weekly sessions, participants will also work to improve coping abilities on their own.
  Arms: 3
Behavioral: Telephone-administered supportive-expressive therapy — Telephone-administered supportive-expressive therapy is aimed to improve relationships with friends, family members, and health care providers. Participants in will partake in 12 weekly conference calls lasting approximately 90 minutes each. Six to eight participants and two group facilitators will be connected via telephone each week. Separate conference call groups will be conducted for men who have sex with men, heterosexual men, and women. The first 60 minutes of each session will focus on discussing topics believed to be of interest to older adults with HIV and providing up-to-date information related to living with HIV/AIDS. The last 30 minutes of each session will be devoted to discussing topics raised by the group.
  Arms: 2
Behavioral: Individual therapy — Participants will receive no active treatment, but will have access to community-based support services that are commonly available to people living with HIV/AIDS. Additionally, participants who experience pronounced periods of emotional crisis and request assistance will be provided with brief, individual, telephone-based therapy by study clinicians.
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of a telephone-delivered coping improvement group intervention in improving quality of life in older adults with HIV.

DETAILED DESCRIPTION:
According to a 2004 report by the Centers for Disease Control and Prevention (CDC), by December, 2003, more than 57,000 people in the United States were 55 years of age or older when they were diagnosed with AIDS. Furthermore, the CDC predicts that, by 2015, 50% of all cases of HIV/AIDS in the U.S. will occur in people 50 years of age or over. HIV infected older adults tend to experience elevated levels of depression and suicidal ideation, confront complex barriers to medical and mental health services, and lack social support resources. Unfortunately, very few interventions are available to improve quality of life in older adults living with HIV/AIDS. Moreover, many older adults with HIV/AIDS do not receive adequate treatment because of geographic isolation, physical limitations, or confidentiality concerns. A therapy program administered via the telephone may be a more accessible option for this population. This study will evaluate the effectiveness of a telephone-delivered coping improvement group intervention in improving quality of life in older adults with HIV.

Participants in this 11-month, single-blind study will first complete self-administered surveys in the privacy of their own homes. Participants will then be randomly assigned to one of the following three study groups: (1) individual therapy upon request; (2) telephone-administered supportive-expressive group therapy; or (3) telephone-administered coping improvement group therapy. Participants in Group 1 will receive no active treatment, but will have access to community-based support services that are commonly available to people living with HIV/AIDS. Additionally, participants in Group 1 who experience pronounced periods of emotional crisis and request assistance will be provided with brief, individual, telephone-based therapy by study clinicians. Participants in Groups 2 and 3 will partake in 12 weekly conference calls lasting approximately 90 minutes each. Six to eight participants and two group facilitators will be connected via telephone each week. Separate conference call groups will be conducted for men who have sex with men, heterosexual men, and women. For Group 2, the first 60 minutes of each session will focus on discussing topics believed to be of interest to older adults with HIV and providing up-to-date information related to living with HIV/AIDS. The last 30 minutes of each session will be devoted to discussing topics raised by the group. For Group 3, cognitive-behavioral principles will be used to evaluate stressor severity, develop problem- and emotion-focused coping skills, determine the relationship between coping strategies and stressor controllability, and optimize coping through use of social support resources. Between weekly sessions, participants will also work to improve coping abilities on their own. All participants will complete follow-up assessments via telephone over the 8 months following completion of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Currently living with HIV or AIDS
* Score of 75 or higher on the Mini-Mental Status Examination

Exclusion Criteria:

* Active use of drugs and/or alcohol
* Poor cognitive functioning

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2007-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Depression | Measured at pre-intervention, post-intervention, and 4- and 8-month follow-up

SECONDARY OUTCOMES:
Coping | Measured at pre-intervention, post-intervention, and 4- and 8-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Cale, Study Chair — Ohio University IRB
Locations (1):
- Ohio University College of Osteopathic Medicine; Geriatric Medicine, Athens, Ohio, United States

REFERENCES:
- [Derived] Heckman BD, Lovejoy TI, Heckman TG, Anderson T, Grimes T, Sutton M, Bianco JA. The moderating role of sexual identity in group teletherapy for adults aging with HIV. Behav Med. 2014;40(3):134-42. doi: 10.1080/08964289.2014.925417. PMID 25090366
- [Derived] Heckman TG, Heckman BD, Anderson T, Lovejoy TI, Mohr D, Sutton M, Bianco JA, Gau JT. Supportive-expressive and coping group teletherapies for HIV-infected older adults: a randomized clinical trial. AIDS Behav. 2013 Nov;17(9):3034-44. doi: 10.1007/s10461-013-0441-0. PMID 23474642
- [Derived] Heckman TG, Sikkema KJ, Hansen N, Kochman A, Heh V, Neufeld S; AIDS and Aging Research Group. A randomized clinical trial of a coping improvement group intervention for HIV-infected older adults. J Behav Med. 2011 Apr;34(2):102-11. doi: 10.1007/s10865-010-9292-6. Epub 2010 Sep 21. PMID 20857188